CLINICAL TRIAL: NCT07394686
Title: Association Between Ultrasonographic Subglottic Airway Measurements and Postoperative Respiratory Adverse Events in Children Under Three Years of Age
Brief Title: Ultrasonographic Subglottic Airway Measurements and Postoperative Respiratory Events in Young Children
Status: Not yet recruiting | Type: Observational
Sponsor: Bursa Sevket Yilmaz Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gürcan Güler, Principal Investigator, Bursa Sevket Yilmaz Training and Research Hospital
Other Study IDs: 2024-TBEK 2025/12-01
Record Dates: First submitted 2026-01-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Perioperative Respiratory Adverse Events; Postoperative Respiratory Complications
Keywords: Postoperative Respiratory Complications; Pediatric airway; Pediatric airway evaluation; Subglottic airway measurements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients under three years of age: This cohort includes children under three years of age undergoing elective surgery. As part of routine perioperative care, ultrasonographic measurements of the subglottic airway are performed during surgery. Participants are followed postoperatively for the occurrence of respiratory-related adverse events.
  Interventions: Other: Ultrasonographic subglottic airway measurement

INTERVENTIONS:
Other: Ultrasonographic subglottic airway measurement — Non-invasive ultrasonographic measurement of the subglottic airway performed intraoperatively as part of routine clinical care. No therapeutic intervention is applied.

SUMMARY:
This study aims to better understand postoperative respiratory adverse events that may occur in some children under three years of age undergoing airway management during surgery. As part of the study, ultrasonographic measurements of a portion of the upper airway will be performed during surgery using a non-invasive ultrasound device. These measurements will be evaluated in relation to perioperative respiratory outcomes. The results of this study may contribute to improved understanding of airway-related factors associated with postoperative respiratory safety in young children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0 to 35 months
* Scheduled for elective surgery under general anesthesia
* Planned airway management with a laryngeal mask airway
* Ability to perform intraoperative ultrasonographic subglottic airway measurements
* Written informed consent obtained from a parent or legal guardian

Exclusion Criteria:

* Known congenital or acquired airway anomalies
* Craniofacial anomalies
* Emergency surgical procedures
* Planned tracheal intubation instead of laryngeal mask airway
* Inability to obtain adequate ultrasonographic subglottic airway measurements

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of children under three years of age scheduled for elective surgery under general anesthesia. All participants undergo planned airway management with a laryngeal mask airway and intraoperative ultrasonographic assessment of the subglottic airway as part of routine clinical care. Written informed consent is obtained from a parent or legal guardian prior to participation.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Perioperative respiratory adverse events (PRAE) | immediately after the surgery
  The occurrence of clinically significant perioperative respiratory adverse events, defined as moderate to severe stridor and/or laryngospasm requiring clinical intervention, including positive pressur

SECONDARY OUTCOMES:
Ultrasonographic subglottic airway dimensions and area | During surgery
  Subglottic airway mediolateral and anteroposterior diameters and the calculated subglottic cross-sectional area measured using ultrasonography at predefined intraoperative time points (T0, T1, and T2). Changes in subglottic airway area between time points (T0-T1, T1-T2, and T0-T2) will also be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Principal Investigator, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sayan O, Erbas M, Sayan M. Association of postoperative airway complications with ultrasonographic measurements in pediatric patients: An exploratory analysis. Saudi J Anaesth. 2025 Oct-Dec;19(4):535-545. doi: 10.4103/sja.sja_215_25. Epub 2025 Sep 3. PMID 40994506
- [Result] Altun D, Sungur MO, Ali A, Bingul ES, Seyhan TO, Camci E. Ultrasonographic Measurement of Subglottic Diameter for Paediatric Cuffed Endotracheal Tube Size Selection: Feasibility Report. Turk J Anaesthesiol Reanim. 2016 Dec;44(6):301-305. doi: 10.5152/TJAR.2016.60420. Epub 2016 Dec 1. PMID 28058141